CLINICAL TRIAL: NCT04246827
Title: Rheumatoid Arthritis Coping Enhancement
Acronym: EMBRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American College of Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00017695
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis; Obesity; Pain
Keywords: rheumatoid arthritis; pain; obesity
MeSH Terms: conditions — Arthritis, Rheumatoid; Obesity; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Lifestyle Weight Management Condition (Experimental): The Enhanced Lifestyle Weight Management condition participants participated in a 12-week protocol in which training in coping skills to increase self-efficacy and decrease the impact of RA pain on behavioral (e.g., activity, eating) and psychosocial (e.g., mood, relationships) weight loss factors was integrated into a lifestyle behavioral weight loss intervention.
  Interventions: Behavioral: Enhanced Lifestyle Weight Management
- Standard Care Control (No Intervention): Participants received standard care of rheumatoid arthritis.

INTERVENTIONS:
Behavioral: Enhanced Lifestyle Weight Management — The Enhanced Lifestyle Weight Management program was a 12-week protocol in which training in coping skills to increase self-efficacy and decrease the impact of RA pain on behavioral (e.g., activity, eating) and psychosocial (e.g., mood, relationships) weight loss factors were integrated into a lifestyle behavioral weight loss intervention.
  Arms: Enhanced Lifestyle Weight Management Condition

SUMMARY:
This study will test an enhanced lifestyle behavioral weight management program that integrates pain coping strategies with a lifestyle intervention that we expect to enhance obese RA patient's ability to cope with pain-related weight challenges. In the proposed study, up to 120 obese (RA-BMI > 28) rheumatoid arthritis patients will be consented in order to randomly assign 80 patients to one of two conditions: 1) an Enhanced Lifestyle Weight Management protocol or 2) standard care control. Patients randomized to the Enhanced Lifestyle Weight Management condition will participate in a 12-week protocol in which training in coping skills to increase self-efficacy and decrease the impact of RA pain on behavioral (e.g., activity, eating) and psychosocial (e.g., mood, relationships) weight loss factors will be integrated into a lifestyle behavioral weight loss intervention.

ELIGIBILITY:
Inclusion Criteria:

* had RA for at least one year
* were 18 to 85 years of age
* were obese according to established RA obesity criteria (RA-BMI > 28)
* had experienced RA pain in the last two weeks.

Exclusion Criteria:

* Subjects were excluded if they 1) have a significant rheumatic disorder other than RA or another organic disease that would significantly affect functioning (e.g., COPD, cancer)
* had a significant medical condition that would expose them to increased risk of a significantly adverse experience during the course of the study (e.g., a recent myocardial infarction)
* they were already involved in a regular exercise program and/or pain coping skills training program
* they had an abnormal cardiac response to exercise such as exercise-induced VT, abnormal blood pressure response, etc.,
* are pregnant at enrollment or at the initiation of intervention
* are younger than 18 years of age or older than 85 years of age
* are known or judged by the physician to be cognitively impaired (dementia, retardation, psychosis)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07-07 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
Change in weight | baseline and post-treatment (12-weeks later)
  Participants' weight was obtained.
Change in waist circumference | baseline and post-treatment (12-weeks later)
  Participants' waist circumference was measured with a standard measuring tape.
Change in body mass index | baseline and post-treatment (12-weeks later)
  Participants' body mass index was calculated by dividing weight (in kg) by height (in m2)
Change in pain as measured by the Brief Pain Inventory | baseline and post-treatment (12-weeks later)
  Pain was assessed with the Brief Pain Inventory, which includes four items asking subjects to rate their usual, worst, least, and average pain during the last week. For each item, patients rate their pain using a scale ranging from 1 to 10 with 1 representing "no pain" and 10 representing "pain as bad as you can imagine."
Change in Physical Disability | baseline and post-treatment (12-weeks later)
  Participants completed the physical functioning scales of the revised Arthritis Impact Scales (AIMS-2). The AIMS-2 assesses the health status of arthritis patients. Scores range from 0 to 10 with 10 representing reduced physical functioning.
Change in Psychological Disability | baseline and post-treatment (12-weeks later)
  Participants completed the psychological functioning scale of the revised Arthritis Impact Scales (AIMS-2). The AIMS-2 assesses the health status of arthritis patients. Scores range from 0 to 10 with 10 representing reduced physical functioning.
Change in C-Reactive Protein | baseline and post-treatment (12-weeks later)
  Serum samples were collected for CRP analysis. All blood specimens were collected in the morning and prior to exercise, centrifuged at 3500 rpm for 10 minutes, and serum stored at -80 degrees Celsius until analysis. CRP is an index of inflammation and activity in RA and is thought to be a more specific measure than erythrocyte sedimentation rate.
Change in Cyclic citrullinated peptide (CCP) antibody | baseline and post-treatment (12-weeks later)
  Cyclic cirtrullinated peptide (CCP) antibody test that is increasingly being used to measure rheumatoid arthritis disease activity, was collected from the eBrowser when available.

SECONDARY OUTCOMES:
Change in physical disability | baseline and post-treatment (12-weeks later)
  The 6 minute walk test was used as an objective assessment of physical disability. This was performed indoors in our lab space, along a long, flat, straight, enclosed corridor. A starting line which marks the beginning and end of each lap was marked on the floor with a brightly colored tape.
Change in rheumatologist Pain Assessment | baseline and post-treatment (12-weeks later)
  The study rheumatologist completed a visual analog scale (VAS) for pain assessment. The VAS was a horizontal line 100 mm in length with anchors ranging from 0 "no disease activity" to 100 "high disease activity."
Change in joint symptoms | baseline and post-treatment (12-weeks later)
  Two joint counts-of tenderness to palpation and of swelling-were obtained by the examining rheumatologist. As suggested by Fuchs and Pincus, we used a reduced count of 28 joints, and counts rather than grading of tenderness and swelling were made, as advocated by Felson et al. (29), to increase inter-observer reliability.
Change in grip strength | baseline and post-treatment (12-weeks later)
  Grip strength was assessed using a sphygmomanometer bulb specially designed for this purpose. Three trials with each hand were conducted, with the average of the three being the person's score.
Change in medication use | baseline and post-treatment (12-weeks later)
  A structured interview was carried out by the study rheumatologist at each evaluation to assess subjects' intake of medication. Subjects were asked what medications they have taken in the two weeks prior to the evaluation. Changes in intake of five categories of medication were scored by comparing data with that collected prior to treatment. The categories included will be 1) nonsteroidal anti-inflammatory drugs, 2) non-narcotic analgesics, 3) narcotics, 4) steroids, and 5) disease modifying anti-rheumatic drugs. Changes in medication were scored as dose increased, dose unchanged, or dose decreased. Based on prior research, we do not anticipate significant changes in medication to occur over the course of the study.

OTHER OUTCOMES:
Change in Arthritis Self-Efficacy Scale (ASES) | baseline and post-treatment (12-weeks later)
  The Arthritis Self-Efficacy Scale (ASES) was used to assess subjects' perceived abilities to perform behaviors that would control arthritis pain and minimize disability. The ASES is a widely used instrument and has been shown to be reliable and valid. Responses for each item range from 10 to 100 where 10 is "very uncertain" and 100 is "very certain."
Change in self-efficacy for weight control | baseline and post-treatment (12-weeks later)
  The Weight Efficacy Life-Style Questionnaire (WEL) is a 20-item scale used to assess subjects' perceived ability to control their weight by resisting eating across five situations (i.e., positive emotions, negative emotions, food availability, social context, physical discomfort). The WEL has demonstrated good reliability and validity. The 20-item measure asks participants to provide information about how certian they are that they can resist overeating across five situations. Response choices range from 0="not at all confident" to 9= "very confident."
Change in Pain Catastrophizing | baseline and post-treatment (12-weeks later)
  Pain catastrophizing was measured using the 13-item Pain Catastrophizing Scale (PCS). This scale measures subjects' tendencies to ruminate about pain, magnify pain, and feel helpless about pain. Participants are provided with a list of thoughts and feelings about pain and are asked to rate the degree to which they have these thoughts/feelings on a scale from 0=not at all to 4=all the time.
Change in Physical activity | baseline and post-treatment (12-weeks later)
  The International Physical Activity Questionnaire (IPAQ) was used to assess change in physical activity. The IPAQ is a short assessment tool that is widely used in adult populations with chronic conditions that asks about individuals' engagement in vigorous, moderate, walking, and sedentary activity over the last 7 days.
Change in eating behavior. | baseline and post-treatment (12-weeks later)
  Tendencies to overeat or binge eat was measured with the Binge Eating Scale (BES). This is a self-report, 16-item questionnaire with multiple choice statements assessing how severely a person overeats. Weights are assigned to each response option ranging from 0 to 3. Higher scores indicate greater severity of over eating.
Change in Mood | baseline and post-treatment (12-weeks later)
  Mood changes were assessed with the condensed version of the Profile of Mood States-B (POMS). This measure uses nine adjective to assess negative and positive mood states.
Change in relationship satisfaction | baseline and post-treatment (12-weeks later)
  Relationship satisfaction was measured with the Interpersonal Support Evaluations List - Short Form (ISEL-SF). This measure includes 16 items that assess perceived support from significant others in these areas: 1) availability of someone to talk to about problems, 2) tangible or instrumental support, 3) belonging support, people available to do things with, and 4) self-esteem support.
Change caloric intake | baseline and post-treatment (12-weeks later)
  Daily food diaries were collected for four consecutive days following each assessment. Participants were sent home with a structured paper diary and asked to record all caloric intake (food and drink) over the four days. Participants were given instructions on how to record their food and will be instructed to contact study staff if they have any questions during the days they are recording their food.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Keefe, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Somers TJ, Wren AA, Blumenthal JA, Caldwell D, Huffman KM, Keefe FJ. Pain, physical functioning, and overeating in obese rheumatoid arthritis patients: do thoughts about pain and eating matter? J Clin Rheumatol. 2014 Aug;20(5):244-50. doi: 10.1097/RHU.0000000000000124. PMID 25036564
- [Derived] Somers TJ, Blumenthal JA, Dorfman CS, Huffman KM, Edmond SN, Miller SN, Wren AA, Caldwell D, Keefe FJ. Effects of a Weight and Pain Management Program in Patients With Rheumatoid Arthritis With Obesity: A Randomized Controlled Pilot Investigation. J Clin Rheumatol. 2022 Jan 1;28(1):7-13. doi: 10.1097/RHU.0000000000001793. PMID 34670994